CLINICAL TRIAL: NCT04855721
Title: A Phase II, Multicenter, Double-blind, Double-dummy, Placebo Controlled, Randomized Study to Evaluate the Efficacy and Safety of AUR101 in Patients With Moderate-to-Severe Psoriasis (INDUS-3)
Brief Title: A Dose-Ranging Phase II Study of AUR101 in Psoriasis (INDUS-3)
Acronym: INDUS-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aurigene Discovery Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUR101-202
Record Dates: First submitted 2021-04-15; First posted 2021-04-22 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Plaque Psoriasis
Keywords: psoriasis; AUR101; ROR; RORgamma; RORgamma inverse agonist; RORgamma inhibitor
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: There are 4 groups in the study; 1 with placebo and 3 with different AUR101 dosing regimens
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, double-dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AUR101 400 mg PO BID (Experimental): Patients will receive AUR101 / placebo in double blind, double dummy manner
  Interventions: Drug: AUR101
- AUR101 200 mg PO BID (Experimental): Patients will receive AUR101 / placebo in double blind, double dummy manner
  Interventions: Drug: AUR101
- AUR101 400 mg PO QD (Experimental): Patients will receive AUR101 / placebo in double blind, double dummy manner
  Interventions: Drug: AUR101
- Placebo (Placebo Comparator): Patients will receive AUR101 / placebo in double blind, double dummy manner
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AUR101 — Oral ROR-gamma inverse agonist
  Arms: AUR101 200 mg PO BID; AUR101 400 mg PO BID; AUR101 400 mg PO QD
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Phase II, Multicenter, Double-blind, Double-dummy, Placebo controlled, Randomized Study to Evaluate the Efficacy and Safety of AUR101 in patients with Moderate-to-Severe Psoriasis (INDUS-3)

DETAILED DESCRIPTION:
This will be a multicenter, double-blind, double-dummy, placebo controlled, randomized study to evaluate the efficacy and safety of AUR101 in patients with moderate-to-severe psoriasis.

Approximately 128 patients with chronic moderate-to-severe plaque psoriasis (defined as Psoriasis Area and Severity Index (PASI) ≥12 and Body Surface Area (BSA) involved ≥10%) will be randomized to four groups (three dose groups of AUR101 and one placebo group) in the ratio of 1:1:1:1.

The patients in each arm will receive AUR101 of 200 mg twice daily, 400 mg twice daily, 400 mg once daily or matching placebo for 16 weeks in a double blind, double dummy fashion. All patients will be followed up for 14 ± 2 days of their last dose for safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of chronic plaque-type psoriasis, diagnosed at least 6 months before screening
2. Psoriasis of at least moderate severity, defined as PASI≥12 and involved BSA≥10 % at screening and Day 1
3. Static 5-point IGA modified [mod] 2011 scale of 3 or higher at screening and Day 1
4. Adult males or females, ≥ 18 to ≤ 70 years of age
5. Ability to communicate well with the investigator and to comply with the requirements of the entire study
6. Willingness to give written informed consent (prior to any study related procedures being performed) and ability to adhere to the study restrictions and assessments schedule

Exclusion Criteria:

1. History of erythrodermic, guttate or pustular psoriasis within last 12 months
2. BMI < 18 or > 40
3. History of lack of response to ustekinumab, secukinumab or ixekizumab (or any therapeutic agent targeted to IL12, IL-17 or IL-23) at approved doses after at least 3 months of therapy
4. Current treatment or history of treatment for psoriasis with any investigational or approved IL-17, IL-12 or IL-23 antagonist biological agents (e.g. secukinumab, briakinumab, tildrakizumab, ustekinumab etc.) within 6 months prior to the first administration of study drug.
5. Current treatment or history of treatment for psoriasis with other investigational or approved biological agents (e.g. anti-TNFα inhibitors - adalimumab, etanercept, infliximab, alefacept etc.) within 3 months prior to the first administration of study drug
6. Current treatment or history of treatment for psoriasis with non-biological systemic medications or immunomodulators (including systemic steroids, apremilast, methotrexate, cyclosporine, acitretin, etc.) or phototherapy within 4 weeks prior to the first administration of study drug.
7. Treatment with medicated topical agents (having active pharmaceutical ingredient that can impact or interfere with the effect of the study drug) within 2 weeks prior to the first administration of study drug.
8. Evidence of organ dysfunction (e.g. liver dysfunction ≥ 1.5 X of ULN for ALT, AST or ALP or Total Bilirubin, or renal dysfunction of ≥ 1.5X of ULN of serum creatinine)
9. Any surgery requiring general anesthesia within 3 months prior to screening
10. History of malignancy within last 5 years except patients with non-melanoma skin cancer or carcinoma in situ of cervix who can participate in the study. Adequately treated cutaneous basal or squamous cell carcinoma are allowed.
11. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV Ab) at screening
12. Patient with known history of systemic tuberculosis or currently suspected or known to have active tuberculosis
13. Patient expected to be started on anti-tubercular therapy either for treatment or prophylaxis of tuberculosis
14. Suspected tuberculosis infection as evident from a positive QuantiFERON TB-Gold test (QFT) or Mantoux test (MT) at screening. Patients with a positive QFT or MT may participate in the study if further work up as per the opinion of the investigator (like Chest X-ray or CT scan of Chest or other locally acceptable method for diagnosing active tuberculosis) establishes that patient does not have active tuberculosis. Patients with latent tuberculosis should not be enrolled except when they are not planned to start prophylaxis for tuberculosis during the study period.
15. History of hypersensitivity or idiosyncratic reaction to any investigational ROR-gamma inhibitors or any of the excipients of study drug
16. History of alcohol or substance abuse that will affect compliance to study procedures/schedule as per Investigator opinion
17. Any previous gastrointestinal surgery or recent (within 3 months) / current history of gastrointestinal disease, that in the opinion of investigator, could impact the absorption of the study drug
18. Positive pregnancy test for women of child-bearing potential (WOCBP) at the screening or randomization visit
19. Male patients who are sexually active with WOCBP, not willing to use reliable contraception methods as mentioned in section 8.14
20. Lactating women or WOCBP who are neither surgically sterilized nor willing to use reliable contraceptive methods (hormonal contraceptive, IUD or any double combination of male or female condom, spermicidal gel, diaphragm, sponge, cervical cap). Please see section 8.14 for acceptable contraceptive practices
21. Has received any investigational biologic agents within 3 months or 5 half-lives (whichever is longer) prior to the first administration of study drug
22. Has received another new chemical entity/non-biologic investigational drug within 28 days or 5 half-lives of investigational drug (whichever is longer) prior to study day 1
23. History of other auto-immune disorders (except psoriasis and psoriatic arthritis) where treatment with systemic immunosuppressants is required
24. History of active infection and/or febrile illness within 7 days prior to Day 1. The infection adequately treated by antibiotics during the screening period as per investigator opinion will be allowed to undergo randomization, provided patient is stable for at least 7 days before randomization
25. Current swab-positive or suspected (under investigation) Covid-19 infection or fever and other signs or symptoms suggestive of Covid-19 infection with recent contact of person(s) with confirmed Covid-19 infection, at screening or Day 1
26. History or presence of any major medical illness (e.g. renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, immunologic, or local active infection/infectious illness) or psychiatric disease, or clinically significant laboratory / ECG abnormalities at screening, any or a combination of illnesses, which, in the opinion of the PI, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study
27. History of any unstable cardiac (including Class III or IV congestive heart failure by New York Heart Association Criteria), respiratory, hepatic, renal or other systemic conditions within 3 months prior to first study drug administration
28. Use of herbal remedies, mega dose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of study drug
29. Patients who have received live attenuated vaccine in the 4 weeks prior to the first administration of study drug -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving PASI 75 response (i.e. 75 percent reduction from baseline PASI [Psoriasis Area and Severity Index] score) at the end of week 12. | Week 12
  PASI-75; A higher proportion of patients reaching PASI-75 means betterment in higher proportion of patients

SECONDARY OUTCOMES:
Proportion of patients achieving PASI 75 response (i.e. 75 percent reduction from baseline PASI [Psoriasis Area and Severity Index] score) at the end of week 4 and 8 | Week 4 and Week 8
  PASI-75; A higher proportion of patients reaching PASI-75 means betterment in higher proportion of patients
Proportion of patients achieving PASI 50, PASI 90 and PASI 100 response at week 12. | Week 12
  PASI-50, PASI-90, PASI-100; A higher proportion of patients reaching PASI-50, PASI-90 or PASI-100 means betterment in higher proportion of patients
Proportion of patients achieving IGA 0 or 1 at week 12 | Week 12
  IGA (Investigator's Global Assessment); Lower scores are better
Percent change from baseline in PASI score at week 12 | Week 12
  Percent Change in PASI from baseline
Percent change from baseline to week 12 in percent BSA involved | Week 12
  Percent Change in BSA (body surface area) from baseline
Proportion of patients achieving DLQI score of 0 or 1 at week 12 | Week 12
  DLQI (Dermatology Life Quality Index) Score; Lower scores are better; Maximum score of 30 and minimum of 0
Plasma Pharmacokinetic parameters at week 4 | Week 4
  Cmax (maximum Plasma concentration)
Plasma Pharmacokinetic parameters at week 4 | Week 4
  AUC0-8 (Area Under The Curve for 8 hours) after morning drug administration
Nature and incidence of Treatment Emergent Adverse Events (TEAEs) | From Day 1 through Follow Up Visit at Week 14
  All Adverse Events which occur from the administration of study drug
Changes in Blood Pressure | From Day 1 through Follow Up Visit at Week 14
  Both systolic and diastolic Blood Pressure changes during trial will be measured
Changes in Pulse Rate | From Day 1 through Follow Up Visit at Week 14
  Pulse Rate changes during trial
Changes in Temperature | From Day 1 through Follow Up Visit at Week 14
  Body temperature changes during trial
Changes in Respiratory Rate | From Day 1 through Follow Up Visit at Week 14
  Respiratory Rate changes during trial
Changes in PR interval in ECG (Electro Cardio Gram) | Week 14 (Follow Up Visit)
  Changes in PR Interval
Changes in QRS interval in ECG (Electro Cardio Gram) | Week 14 (Follow Up Visit)
  Changes in QRS Interval
Changes in QTc interval in ECG (Electro Cardio Gram) | Week 14 (Follow Up Visit)
  Changes in QTc Interval
Changes in CBC (Complete Blood Count) | From Day 1 through Follow Up Visit at Week 14
  Complete Blood Count (CBC)
Changes in Liver Function Tests | From Day 1 through Follow Up Visit at Week 14
  Liver Function Tests (AST, ALT, Total Bilirubin)
Changes in weight | From Day 1 through Follow Up Visit at Week 14
  Weight (in pounds) will be measured at all visits and change in weight (in pounds) will be presented

OTHER OUTCOMES:
Metabolite of AUR101 identification from plasma collected at week 4 | Week 4
  AUR101 metabolites identification in plasma (currently the metabolites are unidentified and no more details are available)
Metabolite of AUR101 quantification from plasma collected at week 4 | Week 4
  AUR101 metabolites quantification in plasma AUR101 (currently the metabolites are unidentified and no more details are available)
Metabolite of AUR101 identification from urine collected at week 4 | Week 4
  AUR101 metabolites identification in urine (currently the metabolites are unidentified and no more details are available)
Metabolite of AUR101 quantification from urine collected at week 4 | Week 4
  AUR101 metabolites quantification in urine (currently the metabolites are unidentified and no more details are available)
Proportion of patients achieving PASI 75 response | Week 16
  PASI-75; A higher proportion of patients reaching PASI-75 means betterment in higher proportion of patients
Proportion of patients achieving PASI 90 response | Week 16
  PASI-90; A higher proportion of patients reaching PASI-90 means betterment in higher proportion of patients
Proportion of patients achieving PASI 100 response | Week 16
  PASI-100; A higher proportion of patients reaching PASI-100 means betterment in higher proportion of patients
Proportion of patients achieving PASI 50 response | Week 16
  PASI-50; A higher proportion of patients reaching PASI-50 means betterment in higher proportion of patients
Proportion of patients achieving IGA 0 or 1 response | Week 16
  IGA 0 or 1; A higher proportion of patients reaching IGA 0 or 1 means betterment in higher proportion of patients
Proportion of patients achieving DLQI 0 or 1 score | Week 16
  DLQI 0 or 1; A higher proportion of patients reaching DLQI 0 or 1 means betterment in higher proportion of patients
Percent change from baseline in PASI score at week 16 | Week 16
  Percent change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Divyesh Mandavia, MD, Study Director — Aurigene Discovery Technologies Limited
Locations (25):
- United States (25):
  - Johnson Dermatology, Fort Smith, Arkansas
  - Northwest AR Clinical Trials Center, Rogers, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - University Clinical Trials, Inc., San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Unison Clinical Trials, Sherman Oaks, California
  - Moore Clinical Research, Inc., Brandon, Florida
  - Skin Research Institute, Coral Gables, Florida
  - Accel Research Sites - Deland CRU, DeLand, Florida
  - FXM Clinical Research Fort Lauderdale, Fort Lauderdale, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Abys New Generation Research Inc., Hialeah, Florida
  - FXM Clinical Research Miami LLC, Miami, Florida
  - Floridian Reserach, Miami, Florida
  - FXM Clinical Research Miramar LLC, Miramar, Florida
  - Lenus Research & Medical Group, LLC, Sweetwater, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Great Lakes Research Group, Inc, Bay City, Michigan
  - Medisearch Clinical Trials, Saint Joseph, Missouri
  - The Dermatology Specialists, New York, New York
  - Sadick Research Group, New York, New York
  - Paddington Testing Co, Inc, Philadelphia, Pennsylvania
  - Dermatology Treatment & Research Center, Dallas, Texas
  - Center for Clinical Studies Ltd., LLP., Webster, Texas

IPD SHARING:
Plan to Share IPD: No
Only IPD (such as SUSAR) required by FDA and IRBs will be shared with other researchers. Aggregate data will be shared with all researchers.